CLINICAL TRIAL: NCT00638339
Title: Effects Of Invasive And Noninvasive Mechanical Ventilation On Sleep In The Icu
Brief Title: Effects Of Invasive And Noninvasive Mechanical Ventilation On Sleep In The Intensive Care Unit (ICU)
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-8053
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Respiratory Insufficiency; Respiration, Artificial; Sleep Deprivation
Keywords: Respiration, artificial; respiratory insufficiency; noninvasive ventilation; sleep deprivation; intensive care units
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration; Sleep Deprivation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: critically ill patients undergoing invasive mechanical ventilation in medical ICU and CCU
- 2: critically ill patients undergoing noninvasive mechanical ventilation in medical ICU and CCU

SUMMARY:
The purpose of this study is to monitor sleep in patients using breathing machines, because little is known about sleep when patients use masks to help their breathing. We'd like to compare sleep in patients using masks to that in patients with a tube in their throats.

DETAILED DESCRIPTION:
Sleep in critically-ill patients is commonly severely fragmented, and sleep architecture is altered as compared to a healthy person. This abnormal sleep may cause some important adverse psychological and physiological consequences. Noise, light, patient-care activities, pain, or medications are some of the contributing factors to sleep disruption in the ICU. Recent evidence also suggests that invasive mechanical ventilation (IMV) itself may lead to sleep fragmentation in the ICU. Noninvasive ventilation (NIV) is a well-established, relatively new form of ventilation which improves sleep quality or gas exchange in some patients with chronic hypoventilatory disorders. Although sleep may be disrupted due to discomfort from the mask or air leaking during NIV use; intermittent use of NIV may result in better sleep quality between NIV sessions. The effects of NIV on sleep in the acute care setting have not yet been studied.

The purpose of the study is to describe the sleep architecture of a cohort of critically-ill patients using NIV, comparing findings to a reference group of patients using (IMV).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs
* Receiving invasive or noninvasive mechanical ventilation
* Anticipated further ventilation of at least 24-hour duration for IMV and 8 hours/ 24 hours for NIV

Exclusion Criteria:

* Pre-morbid diseases that could interfere with interpretation of sleep monitoring including CNS disorders (strokes, encephalopathic states), dementia, and known sleep disorders
* On home BiPAP or CPAP
* Depressed sensorium as evidence by Glasgow Coma Score < 10, need for continuous sedation with Riker Score < 2 and inability to follow verbal commands for sustained 3 hours
* Presence of head trauma, psychiatric illness (including use of antidepressant medication), anoxic brain injury, drug overdose or uncontrolled seizure disorder
* Severe hemodynamic instability (BP< 90 mmHg despite vasopressor therapy) and sepsis
* Recalcitrant hypoxemia (inability to sustain SaO2 > 88%)
* Considered as unstable by ICU team (hemodynamic instability, acute uncontrolled GI bleeding, acute cardiac ischemia or arrhythmias)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients undergoing invasive or noninvasive mechanical ventilation in medical ICU and CCU at Tufts New England Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
To define sleep characteristics in critically-ill patients receiving mechanical ventilation in medical ICU and coronary care unit (CCU) | During 24-hour monitorization period (after recruitment into the study)

SECONDARY OUTCOMES:
To compare total sleep time and differences in sleep architecture including time spent in different sleep stages and arousals in critically-ill patients receiving mechanical ventilation in medical ICU and CCU | During 24-hour monitorization
To determine sleep patterns during NIV use, correlating sleep with periods of use and air leaking | During 24-hour monitorization
To monitor environmental factors including noise, light and patient care activities, and to associate these with sleep patterns | During 24-hour monitorization
To assess associations of severity of illness and sedation usage with sleep patterns | During 24-hour monitorization period

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Ozsancak, MD, Study Director — Research Fellow; Nicholas S Hill, MD, Principal Investigator — Chair of Pulmonary, Critical Care and Sleep Medicine Division
Locations (1):
- Tufts-New England Medical Center Medical ICU and Coronary Care Unit, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No